CLINICAL TRIAL: NCT02398981
Title: Design and Pilot Implementation of a Web Based Real Time Clinical Decision Support Tool. (Checklist for Early Recognition and Treatment of Acute Illness in Pediatrics. CERTAINp
Brief Title: Implementation of a Web Based Real Time Clinical Decision Support Tool.
Acronym: CERTAINp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Grace M. Arteaga, M.D., PI, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-004429
Record Dates: First submitted 2015-02-13; First posted 2015-03-26 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Critical Illness; Sepsis; Respiratory Failure; Shock; Bleeding
MeSH Terms: conditions — Critical Illness; Sepsis; Respiratory Insufficiency; Shock; Hemorrhage | interventions — Checklist

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baseline (No Intervention): Baseline data collection ( 20 patients per ICU)
- Checklist (Experimental): This study is about training and implementation of best critical care practices in the international ICUs with variable resources facilitated by access to a specifically designed electronic checklist 40 patients per ICU
  Interventions: Other: Clinical decision support tool

INTERVENTIONS:
Other: Clinical decision support tool
  Other Names: Checklist
  Arms: Checklist

SUMMARY:
In the developed world critical illness is routinely treated in an intensive care unit (ICU) by highly specialized physicians, nurses and support staff. This model of intensive care is spreading rapidly to low and middle income countries and as it spreads, challenges and limitations to this model arise. In resource-poor settings, inadequate human resources, training, and equipment all present barriers to safe and effective use of life-saving procedures. The advances in medical informatics and human factors engineering have provided tremendous opportunity for novel and user-friendly clinical decision support (CDS) tools that can be applied in a complex and busy hospital setting. Real-time data feeds and standardized patient care tasks in a simulated acute care environment have been proven to have a significant advantage of a novel interface (compared to a conventional) in reducing provider cognitive load and errors. Currently researchers within the investigator's research group have developed and are pilot testing a simple electronic decision support tool: CERTAIN (Checklist for Early Recognition and Treatment of Acute Illness). This tool has been successfully tested and validated in simulated settings and is being implemented as pilot study in 18 countries. Worldwide infant and early childhood mortality continues to be very high partly due to the inability to recognize and respond aggressively to critical illnesses. Investigators expect that adaptation of the algorithms from CERTAIN has potential to be a powerful tool to improve on the medical care of children in developing countries. Investigators aim in this project is 1) to develop a pediatric adaptation of CERTAIN (CERTAINp) and 2) to implement it into clinical practice in resource-poor settings and evaluate the impact of the tool on the processes and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients (< 18 years) admitted for the first time to the participating PICUs will be included.

Exclusion Criteria:

* Not critically ill, admitted for low risk monitoring, planned PICU admission for routine post operative surveillance for less than 24 hours after uncomplicated surgery, readmission and transfer from outside PICU.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 962 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
ICU and hospital lengths of stay | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  Patient will be followed till they get discharged from hospital for whatever length they stay

SECONDARY OUTCOMES:
Adherence to best critical care practices as measured by composite measures of best practice guidelines. | Participants will be followed for the duration of ICU stay, an expected average of 2 weeks
  Adherence to best practice in initial evaluation and treatment of critically ill medical and surgical patients Appropriate shock resuscitation Appropriate sepsis treatment Appropriate mechanical ventilation Appropriate peptic ulcer, deep vein thrombosis and infectious disease prophylaxis. For example Number of patients managed with 100% compliance with sepsis guidelines ( included in the standard operating procedures)/ Number of eligible patients admitted in the time period .

CONTACTS AND LOCATIONS:
Locations (10):
- China (5):
  - Bao'an Maternity & Child Health Hospital, Shenzhen, Guangdong
  - Chengdu 2nd Hospital, Chengdu, Sichuan
  - Chengdu Women & Children's Central Hospital, Chengdu, Sichuan
  - West China Hospital, Chengdu, Sichuan
  - Shanghai Childrens' Medical Center, Shanghai
- University Hospital of Split, Split, Croatia
- Fiji National University, Samabula, Fiji
- JSS hospital, Mysore, Karnataka, India
- Instituto Nacional de Salud del NiÃ±o, Lima, Peru
- Centre Medical Evangelique-Nyankunde, Nyankunde, Eastern Province, Republic of the Congo